CLINICAL TRIAL: NCT04193007
Title: A Randomized Phase II Trial of Brain Radiotherapy Combined With Targeted Therapy in Patients With Asymptomatic NSCLC Brain Metastasis With Gene Sensitive Mutation
Brief Title: The Role of Brain Radiotherapy in Patients With Asymptomatic Brain Metastasis in the Era of Targeted Therapy for NSCLC
Acronym: BRATR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y-Q201802-009
Record Dates: First submitted 2019-11-13; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Non Small Cell Lung Cancer; Brain Metastases
Keywords: Non Small Cell Lung Cancer; Brain Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Molecular Targeted Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- molecular targeted therapy group (Experimental): Molecular targeted therapy(according to the results of gene detection, targeted drugs were selected, such as EGFR mutation using the first generation of EGFR-TKI,ALK or ROS1 mutation using the first generation of ALK inhibitors)
  Interventions: Drug: molecular targeted therapies
- Brain Radiotherapy and molecular targeted therapy group (Experimental): Brain Radiotherapy (stereotactic radiotherapy was used for 1-3 intracranial lesions, and simultaneous modulated accelerated radiation therapy for Brain(SMART-Brain )was used for more than 3 intracranial lesions);Molecular targeted therapy(according to the results of gene detection, targeted drugs were selected, such as EGFR mutation using the first generation of EGFR-TKI,ALK or ROS1 mutation using the first generation of ALK inhibitors)
  Interventions: Drug: molecular targeted therapies; Radiation: Brain Radiotherapy

INTERVENTIONS:
Drug: molecular targeted therapies — if EGFR mutation is positive, (gefitinib, ecotinib, erlotinib）or ALK/ROS-1 positive（Crizotinib）
  Other Names: Targeted Therapy, Molecular; Therapy, Molecular Targeted; Targeted Molecular Therapies
Radiation: Brain Radiotherapy — SRS was used for 1-3 intracranial lesions, and simultaneous modulated accelerated radiation therapy for Brain(SMART-Brain)was used for more than 3 intracranial lesions
  Other Names: Stereotactic radiotherapy,SRS; simultaneous modulated accelerated radiation therapy for Brain,SMART-Brain
  Arms: Brain Radiotherapy and molecular targeted therapy group

SUMMARY:
Brain metastasis is the most common neurological complication in tumor patients, and lung cancer is the most common tumor with brain metastasis. The prognosis of patients with non-small cell lung cancer with brain metastasis is poor. If not treated, the median survival time was about 1 month, the median survival time for steroid therapy was about 2 to 3 months, and the median survival time for patients receiving whole brain radiotherapy was about 3 to 6 months. Studies have shown that the incidence of brain metastasis is not only related to tumor size, N stage and tumor cell type, but also more likely to occur in NSCLC patients with sensitive gene mutation. With the rapid development of NSCLC molecular targeted therapy and precise radiotherapy, the new main therapeutic methods for NSCLC brain metastasis in recent years include stereotactic radiotherapy for (SRT),. Based on intensity modulated technique, simultaneous modulated accelerated radiation therapy for Brain(SMART-Brain) and molecular targeted therapy were carried out. However, at present, the best treatment choice for NSCLC brain metastasis, especially for asymptomatic brain metastasis patients, is still controversial. The choice and combined application mode of individualized treatment for different patients is still a problem to be explored. Based on the synergistic effect of radiotherapy and molecular targeted therapy on the basis of cell and molecule, The purpose of this study was to prospectively compare the efficacy of radiotherapy combined with targeted therapy and targeted therapy alone in patients with asymptomatic NSCLC brain metastasis with gene sensitive mutations, and subgroup analysis of different molecular targets and mutation sites. It is expected that this study will provide a basis for optimizing the curative effect of patients with NSCLC brain metastasis.

DETAILED DESCRIPTION:
This is a randomized phase II clinical trial. The objective of the study is to assess efficacy and safety of brain radiotherapy combined with targeted therapy and simple targeted therapy in patients with asymptomatic NSCLC brain metastasis with gene sensitive mutation. Patients were randomized with equal allocation to Molecular targeted therapy alone or with brain radiotherapy. Study therapy continued until disease progression, unacceptable adverse event, or withdrawal of consent

ELIGIBILITY:
Inclusion Criteria:

* Histology confirmed that it was non-small cell lung cancer;
* EGFR, ALK or ROS1 gene detection showed sensitive gene mutation, and patients were willing to receive targeted therapy;
* brain MRI confirmed brain metastasis;
* asymptomatic or symptomatic brain metastasis could be controlled by glucocorticoid;
* PS score 0-1;
* no brain radiotherapy or targeted therapy before entering the group;
* there was no history of malignant tumor and no serious medical diseases;
* Laboratory examination: White blood cell count ≥ 4 *10^9/L, neutrophil count ≥ 2.0 *10^9, platelet count ≥ 100 *10^9, hemoglobin ≥ 10 g / L, liver and kidney function and ECG were normal;
* the pregnancy test was negative within 3 days before entering the group, and agreed to use medically effective contraceptives during the experiment;
* sign informed consent form.

Exclusion Criteria:

* Small cell lung cancer was confirmed by pathology;
* other malignant tumors (unless PFS ≥ 3 years, except non-black skin cancer);
* were treated with brain radiotherapy or targeted therapy before;
* those with other potentially serious diseases (congestive heart failure, transmural myocardial infarction, admission with severe acute bacterial or fungal infection, COPD or other respiratory diseases that affect treatment, etc.), Taking into account that the study may exacerbate or fail to control the disease;
* severe immunosuppressive diseases, such as AIDS;
* pregnant women, lactating women or women of childbearing age who do not agree with the use of effective contraception in the trial;
* Intracranial metastasis with obvious symptoms or symptoms that can not be relieved by glucocorticoid alone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free survival,iPFS-LM | Every 6 weeks up to 2 years
  Time from BM diagnosis to the first documentation of intracranial lesion progression or death with documented intracranial progression
Objective Response Rate,ORR | 1 month after treatment
  ORR, proportion of patients with a best overall response of complete response or partial response (CR+PR)

SECONDARY OUTCOMES:
Progress Free Survival rate,PFS | Every 6 weeks up to 2 years
  The period from the start of treatment to the progression or death of a patient
Median Survival Time,MST | Every 6 weeks up to 2 years
  the cumulative survival rate is 0.5, the corresponding survival time means that only 50% of the individuals can live through this time.
adverse events | Every 6 weeks up to 2 years
  Number of patients with adverse events (AEs) as a measure of safety and tolerability

OTHER OUTCOMES:
Overall Survival rate, OS | Every 6 weeks up to 2 years, and then every 3 months up to 5 years
  time from the beginning of study to death due to any cause or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Liu Anwen, Phd, Study Director — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Afiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nayak L, Lee EQ, Wen PY. Epidemiology of brain metastases. Curr Oncol Rep. 2012 Feb;14(1):48-54. doi: 10.1007/s11912-011-0203-y. PMID 22012633
- [Result] Mujoomdar A, Austin JH, Malhotra R, Powell CA, Pearson GD, Shiau MC, Raftopoulos H. Clinical predictors of metastatic disease to the brain from non-small cell lung carcinoma: primary tumor size, cell type, and lymph node metastases. Radiology. 2007 Mar;242(3):882-8. doi: 10.1148/radiol.2423051707. Epub 2007 Jan 17. PMID 17229875
- [Result] Shin DY, Na II, Kim CH, Park S, Baek H, Yang SH. EGFR mutation and brain metastasis in pulmonary adenocarcinomas. J Thorac Oncol. 2014 Feb;9(2):195-9. doi: 10.1097/JTO.0000000000000069. PMID 24419416
- [Result] Khalifa J, Amini A, Popat S, Gaspar LE, Faivre-Finn C; International Association for the Study of Lung Cancer Advanced Radiation Technology Committee. Brain Metastases from NSCLC: Radiation Therapy in the Era of Targeted Therapies. J Thorac Oncol. 2016 Oct;11(10):1627-43. doi: 10.1016/j.jtho.2016.06.002. Epub 2016 Jun 23. PMID 27343440
- [Result] Yang P, Kulig K, Boland JM, Erickson-Johnson MR, Oliveira AM, Wampfler J, Jatoi A, Deschamps C, Marks R, Fortner C, Stoddard S, Nichols F, Molina J, Aubry MC, Tang H, Yi ES. Worse disease-free survival in never-smokers with ALK+ lung adenocarcinoma. J Thorac Oncol. 2012 Jan;7(1):90-7. doi: 10.1097/JTO.0b013e31823c5c32. PMID 22134072
- [Result] Aoyama H, Shirato H, Tago M, Nakagawa K, Toyoda T, Hatano K, Kenjyo M, Oya N, Hirota S, Shioura H, Kunieda E, Inomata T, Hayakawa K, Katoh N, Kobashi G. Stereotactic radiosurgery plus whole-brain radiation therapy vs stereotactic radiosurgery alone for treatment of brain metastases: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2483-91. doi: 10.1001/jama.295.21.2483. PMID 16757720
- [Result] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Result] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710
- [Result] Brown PD, Jaeckle K, Ballman KV, Farace E, Cerhan JH, Anderson SK, Carrero XW, Barker FG 2nd, Deming R, Burri SH, Menard C, Chung C, Stieber VW, Pollock BE, Galanis E, Buckner JC, Asher AL. Effect of Radiosurgery Alone vs Radiosurgery With Whole Brain Radiation Therapy on Cognitive Function in Patients With 1 to 3 Brain Metastases: A Randomized Clinical Trial. JAMA. 2016 Jul 26;316(4):401-409. doi: 10.1001/jama.2016.9839. PMID 27458945
- [Result] Steeg PS, Camphausen KA, Smith QR. Brain metastases as preventive and therapeutic targets. Nat Rev Cancer. 2011 May;11(5):352-63. doi: 10.1038/nrc3053. Epub 2011 Apr 7. PMID 21472002
- [Result] Wu YL, Zhou C, Cheng Y, Lu S, Chen GY, Huang C, Huang YS, Yan HH, Ren S, Liu Y, Yang JJ. Erlotinib as second-line treatment in patients with advanced non-small-cell lung cancer and asymptomatic brain metastases: a phase II study (CTONG-0803). Ann Oncol. 2013 Apr;24(4):993-9. doi: 10.1093/annonc/mds529. Epub 2012 Nov 4. PMID 23129122
- [Result] Iuchi T, Shingyoji M, Sakaida T, Hatano K, Nagano O, Itakura M, Kageyama H, Yokoi S, Hasegawa Y, Kawasaki K, Iizasa T. Phase II trial of gefitinib alone without radiation therapy for Japanese patients with brain metastases from EGFR-mutant lung adenocarcinoma. Lung Cancer. 2013 Nov;82(2):282-7. doi: 10.1016/j.lungcan.2013.08.016. Epub 2013 Aug 28. PMID 24021541
- [Result] Fan Y, Huang Z, Fang L, Miao L, Gong L, Yu H, Yang H, Lei T, Mao W. A phase II study of icotinib and whole-brain radiotherapy in Chinese patients with brain metastases from non-small cell lung cancer. Cancer Chemother Pharmacol. 2015 Sep;76(3):517-23. doi: 10.1007/s00280-015-2760-5. Epub 2015 Jul 7. PMID 26148750
- [Result] Schuler M, Wu YL, Hirsh V, O'Byrne K, Yamamoto N, Mok T, Popat S, Sequist LV, Massey D, Zazulina V, Yang JC. First-Line Afatinib versus Chemotherapy in Patients with Non-Small Cell Lung Cancer and Common Epidermal Growth Factor Receptor Gene Mutations and Brain Metastases. J Thorac Oncol. 2016 Mar;11(3):380-90. doi: 10.1016/j.jtho.2015.11.014. Epub 2016 Jan 25. PMID 26823294
- [Result] Soria JC, Tan DSW, Chiari R, Wu YL, Paz-Ares L, Wolf J, Geater SL, Orlov S, Cortinovis D, Yu CJ, Hochmair M, Cortot AB, Tsai CM, Moro-Sibilot D, Campelo RG, McCulloch T, Sen P, Dugan M, Pantano S, Branle F, Massacesi C, de Castro G Jr. First-line ceritinib versus platinum-based chemotherapy in advanced ALK-rearranged non-small-cell lung cancer (ASCEND-4): a randomised, open-label, phase 3 study. Lancet. 2017 Mar 4;389(10072):917-929. doi: 10.1016/S0140-6736(17)30123-X. Epub 2017 Jan 24. PMID 28126333
- [Result] Paris F, Fuks Z, Kang A, Capodieci P, Juan G, Ehleiter D, Haimovitz-Friedman A, Cordon-Cardo C, Kolesnick R. Endothelial apoptosis as the primary lesion initiating intestinal radiation damage in mice. Science. 2001 Jul 13;293(5528):293-7. doi: 10.1126/science.1060191. PMID 11452123
- [Result] Garcia-Barros M, Paris F, Cordon-Cardo C, Lyden D, Rafii S, Haimovitz-Friedman A, Fuks Z, Kolesnick R. Tumor response to radiotherapy regulated by endothelial cell apoptosis. Science. 2003 May 16;300(5622):1155-9. doi: 10.1126/science.1082504. PMID 12750523